CLINICAL TRIAL: NCT01647438
Title: Translating a Heart Disease Lifestyle Intervention Into the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Namratha Kandula, Dr. Namratha Kandula, MD, MPH, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HL113743-01 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Hyperlipidemia; Hypertension; Pre-diabetes; Diabetes
Keywords: South Asians; Diabetes; Physical Activity; Coronary Heart Disease; Lifestyle
MeSH Terms: conditions — Obesity; Hyperlipidemias; Hypertension; Glucose Intolerance; Diabetes Mellitus; Motor Activity; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Print Health Education (Other): Participants receive print health education materials
  Interventions: Other: Print Health Education
- Lifestyle Intervention (Experimental): Six weekly health education classes and phone counseling.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants will enroll in heart disease prevention group sessions focusing on physical activity, diet, weight, and stress management. Each group will have 6 to 8 participants who will attend 6 weekly, 90 minute group education sessions at Metropolitan Asian Family Services. During each session, participants will watch videos on the day's topic followed by discussion, activities, and assistance in setting realistic goals with attention to physical activity, diet, weight, and stress management. Participants will receive telephone support after each session and up to 12 weeks after they have completed the classes to help reinforce learning objectives.
  Arms: Lifestyle Intervention
Other: Print Health Education — Participants will receive primary care referrals and print health education material about heart disease prevention in the mail.
  Arms: Print Health Education

SUMMARY:
Translating a Heart Disease Lifestyle Intervention in the Community study will evaluate the feasibility and initial effectiveness of a community-based, culturally-targeted, lifestyle intervention to improve the cardiovascular health of underserved South Asian (Indian, Pakistani, Bangladeshi, Nepali, and Sri Lankan) Americans. Participants in this study will be randomly assigned to either a group to receive heart disease prevention classes or to another group where they will receive written materials about heart disease prevention.

DETAILED DESCRIPTION:
South Asian individuals were recruited from a community based organization in Chicago and randomly assigned to the print health education group or the SAHELI intervention.

ELIGIBILITY:
Inclusion Criteria:

* South Asians between 30 and 60 years
* Have at least one CHD risk factor: obesity (body mass index > 25 kg/m2- cutoff for obesity in South Asians), hyperlipidemia, hypertension, pre-diabetes, or diabetes.

Exclusion Criteria:

* Inability to speak English, Hindi, or Urdu
* History of clinically evident CVD (e.g. heart attack, stroke)
* Pregnant, lactating, or planning to become pregnant during the study period
* Conditions that inhibit moderate intensity physical activity
* Systolic blood pressure ≥190 or diastolic blood pressure ≥105; Triglycerides ≥ 400
* Using insulin for diabetes
* Significant medical or psychiatric co-morbidities
* Plans to move out of the area within 2 years
* Family/household member enrolled in study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namratha Kandula, MD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Metropolitan Asian Family Services, Chicago, Illinois

REFERENCES:
- [Derived] Jayaprakash M, Puri-Taneja A, Kandula NR, Bharucha H, Kumar S, Dave SS. Qualitative Process Evaluation of a Community-Based Culturally Tailored Lifestyle Intervention for Underserved South Asians. Health Promot Pract. 2016 Nov;17(6):802-813. doi: 10.1177/1524839916650165. Epub 2016 May 24. PMID 27225217
- [Derived] Kandula NR, Dave S, De Chavez PJ, Bharucha H, Patel Y, Seguil P, Kumar S, Baker DW, Spring B, Siddique J. Translating a heart disease lifestyle intervention into the community: the South Asian Heart Lifestyle Intervention (SAHELI) study; a randomized control trial. BMC Public Health. 2015 Oct 16;15:1064. doi: 10.1186/s12889-015-2401-2. PMID 26475629
- [Derived] Kandula NR, Patel Y, Dave S, Seguil P, Kumar S, Baker DW, Spring B, Siddique J. The South Asian Heart Lifestyle Intervention (SAHELI) study to improve cardiovascular risk factors in a community setting: design and methods. Contemp Clin Trials. 2013 Nov;36(2):479-87. doi: 10.1016/j.cct.2013.09.007. Epub 2013 Sep 21. PMID 24060673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community outreach
Groups:
- Primary Care Referral and Print Health Education: Primary Care Referral and Print Health Education: Participants will receive primary care referrals and print health education material about heart disease prevention in the mail.
Period: Overall Study
Arm/Group | Primary Care Referral and Print Health Education | Lifestyle Intervention
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Referral and Print Health Education | Lifestyle Intervention | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7) | 50 (8) | 50 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity (Minutes/Week)
Description: Change from baseline in minutes per week of physical activity measured by accelerometer at 6-months.
Time Frame: baseline and 6-months
Measure: Mean (Standard Error); unit: min/week
Arm/Group | Primary Care Referral and Print Health Education | Lifestyle Intervention
Number analyzed (Participants) | 32 | 31
min/week | 4 (14) | 10 (15)

2. Primary Outcome: Change in Saturated Fat (% of Daily Kilo-calories From Fat) Intake
Description: Change from baseline in saturated fat (% of daily kilo-calories from fat) intake measured by 24-hour food recall at 6-months
Time Frame: baseline and 6-months
Measure: Mean (Standard Error); unit: percentage of kilocalories
Arm/Group | Primary Care Referral and Print Health Education | Lifestyle Intervention
Number analyzed (Participants) | 32 | 31
percentage of kilocalories | 0.58 (0.51) | 0.37 (0.52)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Primary Care Referral and Print Health Education | Lifestyle Intervention
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No